CLINICAL TRIAL: NCT03479515
Title: Use of Bedside Ultrasound to Monitor Body Composition and Neurodevelopmental Outcomes in Formerly-Premature Toddlers
Brief Title: Ultrasound, Peds Body Composition, and Neurodevelopmental Outcomes
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: PEDS-2018-25847
Record Dates: First submitted 2018-03-12; First posted 2018-03-27 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Prematurity
MeSH Terms: conditions — Premature Birth | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Formerly-Premature Toddlers: Data will be used to create and evaluate predictive equation
  Interventions: Device: Ultrasound

INTERVENTIONS:
Device: Ultrasound — Ultrasound, ADP, bioimpedance measurements

SUMMARY:
The overall objective of the proposal is to evaluate the ability of ultrasound to predict the body composition of toddlers in the outpatient clinical setting and to evaluate the relationship between body composition and neurodevelopment.

DETAILED DESCRIPTION:
The investigators will address the hypothesis in the following Specific Aims:

Specific Aim 1: Validate ultrasound as a method to measure whole body fat mass and fat-free mass in toddlers. Body composition will be assessed using ultrasound measurements and the validated method of air displacement plethysmography (ADP).

Specific Aim 2: Determine the effect of a handheld Force-Measuring Ultrasound Probe on intra- and inter-observer variability in ultrasound measurements. A device which measures the force applied to the ultrasound probe will be used to obtain measurements of muscle and adipose tissue thickness (biceps, abdomen, and quadriceps) in toddlers.

ELIGIBILITY:
Inclusion Criteria:

* toddlers who were ≤ 36 weeks gestational age (GA) at birth who attend the University of Minnesota Masonic Children's Hospital NICU Follow Up Clinic
* written consent obtained from a parent before or at time of visit

Exclusion Criteria:

* toddlers who require medical support that prevents them from having ADP measurements taken
* those with an inability to sit in a supported seat for 5 minutes
* those weighing less than 10 kg

Ages: 2 Years to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Toddlers who were ≤ 36 weeks gestational age (GA) at birth who attend the University of Minnesota Masonic Children's Hospital NICU Follow Up Clinic
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2018-07-20 (Actual); Primary Completion 2023-06-06 (Actual); Study Completion 2023-06-06 (Actual)

PRIMARY OUTCOMES:
Ultrasound Measurements | through study completion, up to 2 years
  Tissue thickness (adipose and muscle) will be measured in cm using the ultrasound probe.

SECONDARY OUTCOMES:
Body Composition Measurements | through study completion, up to 2 years
  Fat and fat-free mass will be measured in kilograms using bioimpedance and air displacement plethysmography.
Neurodevelopmental Status for 2 year olds | through study completion, up to 2 years
  Bayley Scales of Neurodevelopment III will be used to measure neurodevelopmental status at 2 years of age, including cognition, language, and motor scores (composite scoring for each area: Cognitive, 55-145; Language, 47-153; Motor, 46-154).
Neurodevelopmental Status for 3 and 4 year olds | through study completion, up to 2 years
  Weschler Preschool and Primary Scale of Intelligence (WPPSI) at 3 and 4 years of age will be used to measure neurodevelopmental status for toddlers 3, 4, or 5 years of age. Quotient and Composite scores have a mean of 100 and a standard deviation of 15. Subtest scaled scores have a mean of 10 and a standard deviation of 3.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Ramel, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Masonic Children's Hospital, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No